CLINICAL TRIAL: NCT06386510
Title: Can Stimulating the Tongue Help Improve Upper Limb Motor Function and Brain Plasticity in Individuals at the Chronic Stage of a Stroke: a Randomized Controlled Trial
Brief Title: Cranial Nerve Neuromodulation to Improve Arm Function and Brain Plasticity in Stroke
Acronym: CN-NINM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-5517
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Cranial nerve non-invasive neuromodulation; Brain plasticity; Recovery; Strength training; Transcranial magnetic stimulation
MeSH Terms: conditions — Stroke | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: multicentered stratified randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real CN-NINM + UL training group (Experimental): Upper limb strength training program combined to real CN-NINM
  Interventions: Procedure: Strength training; Procedure: Cranial nerve non-invasive neuromodulation
- sham CN-NINM + UL training group (Placebo Comparator): Upper limb strength training program combined to sham CN-NINM
  Interventions: Procedure: Strength training; Procedure: Cranial nerve non-invasive neuromodulation

INTERVENTIONS:
Procedure: Strength training — The strength training program will last 4 weeks (3 X/week, 60 minutes). Using dead weights, the 1RM (i.e. the maximal load that an individual can lift once) will be estimated by the 10RM for the wrist extensors and the elbow and shoulder flexors. The grip muscles of the affected hand will also be trained with a JAMAR® dynamometer. Depending on each participant's intensity training group, training will start at 35%, 50% or 70% of 1RM and will be increased by 5% each week to reach, by week 4, 50%, 65% and 85%, for the low, moderate, and high-intensity group, respectively.
Procedure: Cranial nerve non-invasive neuromodulation — For the first 20 minutes of each training session, CN-NINM will be applied (50 μsec at 150 Hz), using a portable stimulator (Cthulhu Shield, USA) with a network of 18 electrodes, directly on the participants' tongue. The participants will hold the device in place by pressing their tongue upwards and the intensity of the stimulus will be set by each participant to a comfortable level of sensation (experimental group) or set by a trainer to a non-perceivable stimulus (control group).

SUMMARY:
Following a stroke, persistent residual muscle weakness in the upper limb (UL) drastically impacts the individuals' quality of life and level of independence. Training interventions are recommended to promote UL motor recovery, and recent studies have shown that training must be tailored to each individual's recovery potential to maximise training gains. Complementary to training interventions, non-invasive brain stimulation devices (NIBS) can help support the provision of post-stroke care by modulating brain excitability and enhancing recovery. Among NIBS, cranial nerve non-invasive neuromodulation (CN-NINM) is gaining increasing attention in rehabilitation since it can directly and non-invasively stimulate the tongue's cranial nerves. The impulses generated can then reach the motor cortex, induce neuroplastic changes and support recovery. Promising results in various neurological populations have been observed, but in stroke, the efficacy of CN-NINM at improving arm motor recovery and brain plasticity is yet to be determined. This is what the present project intends to address, using a stratified randomized controlled trial, where participants in the chronic phase of a stroke will take part in a 4-week individualized training program of their affected UL in combination with real or sham CN-NINM. Before and after the intervention, participants will undergo clinical and neurophysiological evaluations to thoroughly evaluate CN-NINM-induced changes in UL motor function and associated neuroplastic changes. The proposed study will allow an in-depth evaluation of the effects of CN-NINM for an eventual implementation in clinics and at home to support optimal post-stroke recovery.

DETAILED DESCRIPTION:
Residual muscle weakness in the affected upper limb (UL) has a significant negative impact on the performance of activities of daily living (ADL) of individuals with a stroke. Studies report that the degree of UL weakness is strongly correlated to the level of functioning in ADL, thus affecting the overall level of independence post-stroke.

Motor recovery post-stroke is mainly associated with the central nervous system's ability to reorganize, or neuroplasticity. Neuroplasticity can be assessed with non-invasive transcranial magnetic stimulation (TMS). TMS allows for assessing the excitability of the descending corticospinal pathway, the main motor pathway controlling movements of the limbs and trunk. The amplitude of TMS-elicited motor evoked potentials (MEP) gives a direct measure of the excitability of corticospinal neurons and studies have shown that MEP amplitudes can be used to probe neuroplastic changes associated with motor recovery and are good predictors of an individual response to exercise post-stroke. In a recent study on UL exercises in chronic stroke survivors, baseline MEP amplitudes were used to estimate participants' potential for recovery and to tailor the intensity of the UL training program accordingly. By stratifying them based on their MEP amplitudes, all participants, regardless of their level of post-stroke recovery, showed significant improvements in UL function following their tailored training program. Collectively, these results suggest that assessing MEP amplitude can provide an efficient way to evaluate neuroplasticity as well as to assist in staging and tailoring individuals' training intervention to optimize post-stroke recovery.

To enhance neuroplasticity, training exercises are critical to rehabilitation post-stroke since they allow for improvement in UL motor function and strength as well as promote brain plasticity, leading to increased use of the UL in ADLs. To capitalize on the benefit of strength training at promoting motor recovery and neuroplasticity, non-invasive brain neurostimulation (NIBS) modalities are increasingly studied as an adjunct therapy in stroke rehabilitation. To date, transcranial direct current stimulation (tDCS) is the most studied NIBS, but a great variability in response to tDCS is noted, with more than 50% of individuals not responding as expected. This heterogeneity across studies in tDCS response could be explained by the absence of a consensus on optimal stimulation parameters, the influence of individual brain anatomical characteristics on the response to tDCS and the presence of an electric current shunting through the skull. Thus, to counteract the impact of inter-individual anatomical variability and electrical current shunting by the skull, recent studies are now investigating cranial nerve stimulation as an adjunct therapy in stroke when paired with rehabilitation. An emerging NIBS therapeutic device, stimulating two major cranial nerves, the trigeminal and glossopharyngeal nerves, by tongue stimulation, is making its way into neurological rehabilitation, that is cranial nerve non-invasive neuromodulation (CN-NINM). By applying electrodes directly to the tongue, CN-NINM allows the generation of a direct flow of neural impulses that travel to the cranial nerve nuclei of the brainstem and then to the motor cortex to induce targeted neuroplastic changes when combined with rehabilitation treatments. Following various neurological injuries and combined with many interventions, CN-NINM results in improved functional performance such as walking and balance. Neuroplasticity changes have also been observed such as an increase in the brain beta activation measured with electroencephalography and increased activation in the primary motor cortex area. Post-stroke, only one study has compared the impact of CN-NINM combined with a 2-week balance and gait training program (experimental group) to a 2-week balance and gait training program alone (control group) on functional performance, as assessed with the Mini-Best test, in individuals in the subacute stage of a stroke. Based on Mini-Best test score, an improvement in balance in the experimental group compared with the control group was noted (p=0.032). Although promising, CN-NINM has not been studied to improve UL function, despite the negative impact of UL impairment on post-stroke functional performance. Also, to lay the foundation for the applicability of this NIBS in stroke, understanding the neurophysiological effects of CN-NINM by evaluating neuroplasticity changes is crucial.

Objective: The main objective is to assess the impact of CN-NINM combined with a tailored UL strength training program on improvement in UL function and brain excitability in individuals at the chronic stage of a stroke. The secondary objective is to assess the presence of a relationship between UL functional gain and change in brain excitability for the study sample.

Methods: In this multicentered stratified randomized controlled trial, 74 participants will be recruited and stratified according to the baseline amplitude of their TMS-induced MEP responses into three strata of training intensity: 1) low-intensity (MEP 20-49μV); 2) moderate-intensity (MEP 50-120uV) and 3) high-intensity (MEP>120uV). . Within each stratum, participants will be randomized into the experimental group (real CN-NINM + UL strength training) or the control group (sham CN-NINM + UL strength training). Sociodemographic and stroke-related variables (e.g., age, time since stroke) will be collected to confirm participant eligibility. Prior to and at the end of the intervention, participants will undergo a clinical evaluation of their affected UL as well as a neurophysiological brain evaluation with TMS. The intervention will consist of a 4-week UL strength training program (3X/week, 60-minute duration) combined to a 20-minute CN-NINM application. For the experimental group, the intensity of the stimulus will be set by each participant to a comfortable level of sensation, similar to the sensation in the mouth of a soft drink. For the control group, participants will wear the device such as the experimental group, but the intensity will be controlled by the trainer and set to a non-perceivable stimulus.

ELIGIBILITY:
Inclusion Criteria:

* be ≥18 years of age;
* have had a unilateral supratentorial stroke;
* be in a chronic stage of recovery (>6 months);
* present some UL motor recovery (Fugl-Meyer Stroke Assessment [FMA-UE] score ≥25/66);
* are not involved in rehabilitation treatments.

Exclusion Criteria:

* significant spasticity at UL (score >3 on the modified Ashworth scale);
* major sensory deficit at UL (a score <25/34 on the Nottingham sensory assessment and a score <6 on the vibration threshold assessment);
* hemineglect (> 70% of unshaded lines on the same side as the motor deficit on the Line Cancellation test);
* apraxia (score >2.5 on the Alexander test);
* a neurological disorder other than stroke-related;
* orthopedic problems at UL;
* cognitive impairment (score <2/5 on the Mini-Cog);
* significant pain intensity at UL (a score ≥ 6/10 on the Visual Analog Pain Scale);
* absence of MEP (peak-to-peak MEP amplitude <20μV);
* contraindications to CN-NINM and TMS.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in UL motor function on the Fugl-Meyer Stroke Assessment Scale | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM
  Change in motor function of the affected UL will be assessed using the Fugl-Meyer Stroke Assessment. The score of this scale range from 0 (no motor recovery) to 66 (full motor recovery).
Change in UL functional performance on the Wolf Motor Function Test | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in functional performance of the affected UL will be assessed with the timed score of the Wolf Motor Function Test; comprising 17 tasks. The maximal time allocated to each task is 120 seconds.
Change in motor cortex excitability by means of resting MEP amplitudes elicited by TMS over both hemispheres. | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in motor cortex excitability will be assessed by resting peak-to-peak MEP amplitudes of the affected and unaffected first dorsal interosseous muscles (FDI) at 130% of the FDI resting motor threshold over 20 trials

SECONDARY OUTCOMES:
Change in participants' subjective real life functional UL performance on the Motor Activity Log | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in participants' self-reported affected UL performance in everyday activities will be assessed with the Motor Activity Log (MAL). The MAL comprises 14 task scored on a 0 to 5 Likert scale, where a score of 5 represents normal quantity and quality of use of affected UL.
Change in active and passive range of motion at both UL in shoulder flexion, elbow flexion and wrist extension | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in active and passive range of motion at both UL will be assessed in degrees with a manual goniometer
Change in resting motor threshold of the affected and unaffected FDI | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in resting motor threshold of the affected and unaffected FDI will be assessed with TMS and described as % of output stimulator

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Helene Milot, PhD, Principal Investigator — Université de Sherbrooke
Locations (3):
- Canada (3):
  - CRIR/Feil/Oberfeld Research Center; Centre intégré de santé et de services sociaux de Laval; Jewish Rehabilitation Hospital, Laval, Quebec
  - CIRRIS, Québec, Quebec
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec